CLINICAL TRIAL: NCT03554473
Title: Safety Run-In and Phase II Trial of M7824 and Topotecan or Temozolomide in Relapsed Small Cell Cancers
Brief Title: M7824 and Topotecan or Temozolomide in Relapsed Small Cell Lung Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anish Thomas, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180110; 18-C-0110
Record Dates: First submitted 2018-06-09; First posted 2018-06-13 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Small Cell; Lung Cancer; Small Cell Lung Cancer
Keywords: Chemosensitivity; DNA Damage and Replication; PD-1/PD-L1; Solid Tumors; Checkpoint Inhibitors
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Topotecan; Temozolomide; Electrocardiography; Tomography, X-Ray Computed; Positron-Emission Tomography; Acetaminophen; Histamine Antagonists; Diphenhydramine; Dexamethasone; Calcium Dobesilate; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A/M7824 (MSB0011359C) Monotherapy (Experimental): M7824 (MSB0011359C) intravenous (IV) monotherapy once every 21 days on a 21-day cycle. If patients have progressive disease on arm A, they may receive combination therapy of M7824 and Temozolomide.
  Interventions: Drug: M7824; Drug: Temozolomide; Diagnostic Test: EKG; Diagnostic Test: CT scan; Diagnostic Test: PET scan; Drug: Acetaminophen; Drug: Antihistamines; Drug: Diphenhydramine; Drug: Dexamethasone; Drug: Epinephrine
- Arm B/M7824 (MSB0011359C) Plus Topotecan (Experimental): M7824 (MSB0011359C) intravenous (IV) on day 1 plus topotecan (IV) on days 1-5 of a 21-day cycle. At least 6 subjects to receive M7824 plus topotecan to determine safety. 4 more patients enrolled at initial or lower dose for efficacy. If efficacious, an additional 12 subjects enrolled.
  Interventions: Drug: M7824; Drug: Topotecan; Diagnostic Test: EKG; Diagnostic Test: CT scan; Diagnostic Test: PET scan; Drug: Acetaminophen; Drug: Antihistamines; Drug: Diphenhydramine; Drug: Dexamethasone; Drug: Epinephrine
- Arm C/M7824 (MSB0011359C) Plus Temozolomide (Experimental): M7824 (MSB0011359C) intravenous (IV) days 1 and 15 plus temozolomide (oral) on days 1-5 of a 28-day cycle. At least 6 subjects with small cell lung cancer (SCLC) to receive M7824 plus temozolomide to determine safety. 4 more SCLC patients enrolled at initial or lower dose for efficacy. If efficacious, an additional 12 SCLC subjects enrolled. After the 6 safety SCLC cohort, subjects with extrapulmonary small cell cancers will be enrolled.
  Interventions: Drug: M7824; Drug: Temozolomide; Diagnostic Test: EKG; Diagnostic Test: CT scan; Diagnostic Test: PET scan; Drug: Acetaminophen; Drug: Antihistamines; Drug: Diphenhydramine; Drug: Dexamethasone; Drug: Epinephrine

INTERVENTIONS:
Drug: M7824 — Arm A & B: 2400mg intravenous (IV) over up to 120 minutes every 3 weeks on a 3-week cycle. Arm C: 1200 mg IV over 1 hour every 2 weeks on a 4-week cycle.
  Other Names: MSB0011359C
Drug: Topotecan — Arm B: 1 mg/m(2) intravenous (IV) over 30 minutes days 1-5 on a 3-week cycle.
  Other Names: Hycamtin
  Arms: Arm B/M7824 (MSB0011359C) Plus Topotecan
Drug: Temozolomide — Arm C and progressive disease patients on Arm A: 200 mg/m(2) by mouth (PO) days 1-5 on a 4-week cycle.
  Other Names: Temodar
  Arms: Arm A/M7824 (MSB0011359C) Monotherapy; Arm C/M7824 (MSB0011359C) Plus Temozolomide
Diagnostic Test: EKG — Screening and baseline.
  Other Names: Electrocardiogram
Diagnostic Test: CT scan — Computed tomography (CT) scan performed at Screening and after every 2 cycles (6 weeks) per Study Calendar for Arm B 3.5.2, Arm B 3.5.2, and/or Arm C 3.5.3 as applicable.
  Other Names: Computed tomography scan
Diagnostic Test: PET scan — Positron emission tomography (PET) not mandatory - If a computed tomography (CT) scan is not sufficient to assess response, a PET scan may be added per Study Calendar for Arm A 3.5.1, Arm B 3.5.2, and/or Arm C 3.5.3 as applicable.
  Other Names: Positron emission tomography scan
Drug: Acetaminophen — For infusion related reaction, 500-1000 mg by mouth (PO) prior to infusion.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Antihistamines — As medically indicated.
Drug: Diphenhydramine — For infusion related reaction, 50 mg by mouth (PO) prior to infusion.
  Other Names: Benadryl; Banophen; Nytol
Drug: Dexamethasone — As medically indicated.
  Other Names: Maxidex; Ozurdex; DexPak 10 day
Drug: Epinephrine — As medically indicated.
  Other Names: Adrenaline

SUMMARY:
BACKGROUND:

* Small cell lung cancer (SCLC) is an aggressive cancer with a poor prognosis. Although highly responsive to chemotherapy initially, SCLC relapses quickly and becomes refractory to treatment within a few months.
* The inability to destroy residual SCLC cells despite initial chemosensitivity suggests the existence of a highly effective deoxyribonucleic acid (DNA) damage response network. SCLC is also characterized by high DNA replication stress (retinoblastoma (RB1) inactivation, MYC and CCNE1 activation).
* There is only one Food and Drug Administration (FDA) approved treatment for patients with relapsed SCLC after first-line chemotherapy: topotecan, which inhibits religation of topoisomerase I-mediated single-strand DNA breaks leading to lethal double-strand DNA breaks. Temozolomide, an oral alkylating agent, which causes DNA damage by alkylating guanine at position O6 also has activity in relapsed SCLC, particularly for brain metastases.
* Preliminary evidence indicates that disruption of the immune checkpoint programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) pathway can yield responses in a subset of SCLC patients, but response rates (approximately equal to 10%) are lower than non-small cell lung cancer (NSCLC) and other tumors with comparable tumor mutational burden indicating additional immunosuppressive mechanisms at play in the SCLC tumor microenvironment.
* M7824 (MSB0011359C) is a bifunctional fusion protein consisting of an anti-programmed death ligand 1 (PDL1) antibody and the extracellular domain of transforming growth factor beta (TGF-beta) receptor type 2, a TGF-beta trap.
* Safety data from the dose-escalation study in solid tumors as well as preliminary data from expansion cohorts show that M7824 has a safety profile similar to other checkpoint inhibiting compounds.
* Combining immunotherapy, and chemotherapy could synergistically improve the anticancer activity of immunotherapy. Combination of chemotherapy with immunotherapy have improved outcomes in NSCLC and melanoma leading to Food and Drug Administration (FDA) approvals of such combinations.
* We hypothesize that increased DNA damage induced by topotecan and temozolomide will complement the anti-tumor activity of M7824, in recurrent SCLC.

OBJECTIVE:

- The primary objective of the trial is to determine the efficacy (using objective response rate) of M7824 plus topotecan or temozolomide in relapsed SCLC.

ELIGIBILITY:

* Subjects with histological or cytological confirmation of SCLC.
* Subjects must be greater than or equal to 18 years of age and have a performance status (Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.
* Subjects must not have received chemotherapy or undergone major surgery within 2 weeks and radiotherapy within 24 hours prior to enrollment.
* Subjects must have adequate organ function and measurable disease.

DESIGN:

* Arm A (M7824 monotherapy): Up to 10 patients may be treated with M7824 monotherapy to obtain safety and pharmacokinetic (PK) data, and a preliminary estimate of clinical responses to M7824 in SCLC. Patients with progressive disease on Arm A may then receive M7824 plus temozolomide as per description of treatment for Arm C.
* Arm B (M7824 plus topotecan) and Arm C (M7824 plus temozolomide) will be administered in 3 and 4-week cycles respectively; these arms will have a safety run-in followed by efficacy analysis. Up to 10 patients with extrapulmonary small cell cancer will be enrolled in arm C to receive the combination of M7824 and temozolomide.
* Optional tumor biopsies will be obtained at pre-treatment on cycle 1 day 1 (C1D1) and C1D15 for Arm C; pre-treatment on C1D1 and cycle 2 day 1 (C2D1) for arms A and B.
* Every subject of each arm of the safety run-in will be observed for at least 7 days after first dose of M7824 before the subsequent subject can be treated. Subjects who are not evaluable for dose-limiting toxicity (DLT) will be replaced and not included into evaluation.

ARMS:

* Arm A (3-week cycles): M7824 monotherapy 2400 mg every 3 weeks until disease progression or a criterion in Protocol is met. Patients with progressive disease on Arm A may then receive 1200 mg M7824 every 2 weeks plus temozolomide 200 mg/m^2/day on days 1-5 every 4 weeks.
* Arm B (3-week cycles): M7824 2400 mg plus topotecan 1 mg/m(2) on days 1-5 every 3 weeks until disease progression or a criterion in Protocol is met.
* Arm C (4-week cycles): M7824 1200 mg every 2 weeks plus temozolomide 200 mg/m(2)/day on days 1-5 every 4 weeks until disease progression or a criterion in Protocol is met.

DETAILED DESCRIPTION:
Background

Small cell lung cancer (SCLC) is an aggressive cancer with a poor prognosis. Although highly responsive to chemotherapy initially, SCLC relapses quickly and becomes refractory to treatment within a few months.

Extrapulmonary small cell cancers are extremely rare and management of systemic disease with chemotherapy is patterned after the approach used in SCLC.

The inability to destroy residual SCLC cells despite initial chemosensitivity suggests the existence of a highly effective deoxyribonucleic acid (DNA) damage response network. SCLC is also characterized by high DNA replication stress (retinoblastoma (RB1) inactivation, MYC and CCNE1 activation). Similarly, extrapulmonary small cell cancers have no standard treatments and it appears that although these cancers can arise by different mechanisms, they have in common high replication stress, that may be susceptible to DNA damage and immune checkpoint blockade.

There is only one Food and Drug Administration (FDA) approved treatment for patients with relapsed SCLC after first-line chemotherapy: topotecan, which inhibits religation of topoisomerase I-mediated single-strand DNA breaks leading to lethal double-strand DNA breaks. Temozolomide, an oral alkylating agent, which causes DNA damage by alkylating guanine at position O6 also has activity in relapsed SCLC, particularly for brain metastases.

Preliminary evidence indicates that disruption of the immune checkpoint programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) pathway can yield responses in a subset of SCLC patients, but response rates (approximately 10%) are lower than NSCLC and other tumors with comparable tumor mutational burden indicating additional immunosuppressive mechanisms at play in the SCLC tumor microenvironment.

M7824 (MSB0011359C) is a bifunctional fusion protein consisting of an anti-programmed death ligand 1 (PD-L1) antibody and the extracellular domain of transforming growth factor beta (TGF- beta) receptor type 2, a TGF- beta trap.

Safety data from the dose-escalation study in solid tumors as well as preliminary data from expansion cohorts show that M7824 has a safety profile similar to other checkpoint inhibiting compounds.

Combining immunotherapy, and chemotherapy could synergistically improve the anticancer activity of immunotherapy. Combination of chemotherapy with immunotherapy have improved outcomes in non-small cell lung cancer (NSCLC) and melanoma leading to FDA approvals of such combinations.

We hypothesize that increased DNA damage induced by topotecan and temozolomide will complement the anti-tumor activity of M7824, in recurrent SCLC.

Objective

The primary objective of the trial is to determine the efficacy (using objective response rate) of M7824 plus topotecan or temozolomide in relapsed SCLC.

Eligibility

Subjects with histological or cytological confirmation of SCLC or extrapulmonary small cell cancers.

Subjects must be greater than or equal to 18 years of age and have a performance status Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.

Subjects must not have received chemotherapy or undergone major surgery within 2 weeks and radiotherapy within 24 hours prior to enrollment.

Subjects must have adequate organ function and measurable disease.

Design

Arm A (M7824 monotherapy): Up to 10 patients may be treated with M7824 monotherapy to obtain safety and PK data, and a preliminary estimate of clinical responses to M7824 in SCLC. Patients with progressive disease on Arm A may then receive M7824 plus temozolomide as per description of treatment for Arm C.

Arm B (M7824 plus topotecan) and Arm C (M7824 plus temozolomide) will be administered in 3 and 4-week cycles respectively; these arms will have a safety run-in followed by efficacy analysis. Up to 10 patients with extrapulmonary small cell cancer will be enrolled in arm C to receive the combination of M7824 and temozolomide.

Optional tumor biopsies will be obtained at pre-treatment on cycle 1 day 1 (C1D1) and C1D15 for Arm C; pre-treatment on C1D1 and cycle 2 day 1 (C2D1) for arms A and B.

Every subject of each arm of the safety run-in will be observed for at least 7 days after first dose of M7824 before the subsequent subject can be treated. Subjects who are not evaluable for dose-limiting toxicity (DLT) will be replaced and not included into evaluation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed small cell lung cancer (SCLC) or extrapulmonary small cell cancers.
* Subjects with relapsed SCLC (diagnosed with limited or extensive stage disease) with tumor progression on or after at least one prior chemotherapy. Patients with SCLC should in addition have received and have disease progression on or after prior immunotherapy.
* Male and female subjects greater than or equal to 18 years of age. Because no dosing adverse event data are currently available on the use of topotecan, temozolomide and M7824 in subjects 18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status greater than or equal to 2.
* Subjects must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Subjects must not have received chemotherapy or undergone major surgery within 2 weeks and radiotherapy within 24 hours prior to enrollment.
* Patients must have adequate organ and marrow function as defined below:

  * hemoglobin greater than or equal to 9.0 g/dL
  * absolute neutrophil count greater than or equal to 1.5x109/L
  * platelets greater than or equal to 100x10^9/L
  * total bilirubin less than or equal to 2.0 mg/dL
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 x upper limit of normal (ULN) or if liver metastases were present, less than or equal to 5 x ULN
  * creatinine less than or equal to 1.5 mg/dL

OR

--creatinine clearance greater than or equal to 40 mL/min

* Ability of subject to understand and the willingness to sign a written informed consent document.
* The effects of the trial treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly-effective contraception prior to study entry, for the duration of study participation and up to 6 months for women and 3 months for men after the last dose of study drug. Men should not donate sperm during participation in the study and for up to 3 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Subjects with tumor amenable to potentially curative therapy per principal investigator (PI).
* Subjects who are receiving any other investigational agents. Prior immunotherapy, topotecan and temozolomide are allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to (study agent) or other agents used in study.
* Subjects with symptomatic brain metastases will be excluded from trial secondary to poor prognosis. However, subjects who have asymptomatic brain metastases, and those had treatment for their brain metastasis and whose brain disease is stable without steroid therapy for 2 weeks may be enrolled (replacement doses less than or equal to 10 mg of prednisone or equivalent per day are allowed).
* Subjects with evidence of severe or uncontrolled systemic disease, or any concurrent condition, which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies (human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are eligible), Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 3 months, uncontrolled cardiac arrhythmia, stroke/cerebrovascular accident within the past 3 months, bleeding diathesis or recent (within 3 months) clinically significant bleeding events or psychiatric illness/social situations which would jeopardize compliance with the protocol.
* Pregnant women are excluded from this study because topotecan and temozolomide are Class D agents with the potential for teratogenic or abortifacient effects and because the effects of M7824 on the developing human fetus are currently unknown. In addition, because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with topotecan, temozolomide or M7824, breastfeeding should be discontinued if the mother is treated with these agents
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with the exceptions:

  * Diabetes type I, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible;
  * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses less than or equal to 10 mg of prednisone or equivalent per day;
  * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable.
* Systemic therapy with immunosuppressive agents within 7 days before enrollment.
* Administration of live vaccines within 30 days prior to the first administration of study intervention. Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved Coronavirus Disease (COVID) vaccines are permitted.
* Subjects unwilling to accept blood products as medically indicated.
* Known contraindication for topotecan or temozolomide

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0110.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Relapsed Small Cell Lung Cancers (SCLC). Extrapulmonary Small Cell Cancer (ESCC).
Groups:
- Arm A/M7824 (MSB0011359C) Monotherapy: M7824 (MSB0011359C) intravenous (IV) monotherapy once every 21 days on a 21-day cycle. If patients have progressive disease on arm A, they may receive combination therapy of M7824 and Temozolomide.
  First 7 patients on Arm A received dose of 1800mg intravenous (IV) over 60 minutes
  M7824: Arm A & B: 2400mg intravenous (IV) over up to 120 minutes every 3 weeks on a 3-week cycle. Arm C: 1200 mg IV over 1 hour every 2 weeks on a 4-week cycle.
  Temozolomide: Arm C and progressive disease patients on Arm A: 200 mg/m(2) by mouth (PO) days 1-5 on a 4-week cycle.
- Arm C/M7824 (MSB0011359C) Plus Temozolomide: M7824 (MSB0011359C) intravenous (IV) days 1 and 15 plus temozolomide (oral) on days 1-5 of a 28-day cycle. At least 6 subjects with small cell lung cancer (SCLC) to receive M7824 plus temozolomide to determine safety. 4 more SCLC patients enrolled at initial or lower dose for efficacy. If efficacious, an additional 12 SCLC subjects enrolled. After the 6 safety SCLC cohort, 10 subjects with extrapulmonary small cell cancers will be enrolled.
  M7824: Arm A & B: 2400mg intravenous (IV) over up to 120 minutes every 3 weeks on a 3-week cycle. Arm C: 1200 mg IV over 1 hour every 2 weeks on a 4-week cycle.
  Temozolomide: Arm C and progressive disease patients on Arm A: 200 mg/m(2) by mouth (PO) days 1-5 on a 4-week cycle.
Period: Arm A M7824 Relapsed SCLC
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Started | 13 | 0 | 0
Disease Progression | 10 | 0 | 0
Initial Safety Cohort | 7 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrew for hospice care. | 2 | 0 | 0
Not completed — Worsening brain metastases. Did not complete a full cycle or return for restaging. | 1 | 0 | 0
Period: Arm B M7824 + Topotecan Relapsed SCLC
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Started | 0 | 5 | 0
Initial Safety Cohort | 0 | 0 | 0
Completed | 0 | 5 | 0
Not Completed | 0 | 0 | 0
Period: Arm C M7824 + Temozolomide Relapsed SCLC
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Started | 0 | 0 | 10
Initial Safety Cohort | 0 | 0 | 6
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 0
Period: Arm C M7824 + Temozolomide ESCC
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Started | 0 | 0 | 9
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 4
Not completed — Developed progressive disease during Cycle 1. Did not complete a full cycle or return for restaging. | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm A/M7824 (MSB0011359C) Monotherapy: M7824 (MSB0011359C) intravenous (IV) monotherapy once every 21 days on a 21-day cycle. If patients have progressive disease on arm A, they may receive combination therapy of M7824 and Temozolomide.
  First 7 patients received dose of 1800mg intravenous (IV) over 60 minutes
  M7824: Arm A & B: 2400mg intravenous (IV) over up to 120 minutes every 3 weeks on a 3-week cycle. Arm C: 1200 mg IV over 1 hour every 2 weeks on a 4-week cycle.
  Temozolomide: Arm C and progressive disease patients on Arm A: 200 mg/m(2) by mouth (PO) days 1-5 on a 4-week cycle.
- Total: Total of all reporting groups
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide | Total
Number analyzed (Participants) | 13 | 5 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 12 | 22
  >=65 years | 6 | 2 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.85 (11) | 62.6 (9.71) | 59 (12.45) | 61.54 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7 | 14
  Male | 7 | 4 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 5 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4
  White | 12 | 4 | 14 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 5 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Evaluable Participants Who Experience a Partial Response (PR) or Complete Response (CR) Reported Along With an 80% Confidence Interval.
Description: The fraction of evaluable participants who experience a PR or CR will be determined and this fraction will be reported along with an 80% confidence interval. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete response is disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: 6 weeks (Arm B) or 8 weeks (Arm C)
Population: 7/37 participants were not analyzed because 7 participants were not evaluable for response. They did not complete a full cycle followed by restaging.
Measure: Number (80% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 10 | 5 | 15
Proportion of participants
  Partial Response | 0.1 [0 to 0.2216] | 0 [0 to 0] | 0.2 [0.067 to 0.3324]
  Complete Response | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Proportion of Evaluable Participants Who Experience a Partial Response (PR) or Complete Response (CR) Reported Along With an 95% Confidence Interval.
Description: The fraction of evaluable participants who experience a PR or CR will be determined and this fraction will be reported along with an 95% confidence interval. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete response is disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: 6 weeks (Arm B) or 8 weeks (Arm C)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 10 | 5 | 15
Proportion of participants
  Partial Response | 0.1 [0 to 0.2859] | 0 [0 to 0] | 0.2 [0 to 0.4024]
  Complete Response | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: Number of Participants Experiencing a Dose-limiting Toxicity (DLT) by Grade and Type
Description: Fraction of participants experiencing a dose-limiting toxicity (DLT) by grade and type assessed by the CTCAE. Grade 3 is severe. Grade 4 is life threatening. Grade 5 is death related to adverse event. The occurrence of any of the following toxicities will be considered a DLT if judged by the Investigator to be possibly, probably or definitely related to study drug administration: Grade 4 non-hematologic toxicity (not laboratory). Grade 4 hematologic toxicity lasting ≥7 days. Grade 3 non-hematologic toxicity (not laboratory, specifically nausea, vomiting and diarrhea) lasting >5 days despite optimal supportive care. Febrile neutropenia Grade 3 or Grade 4. Thrombocytopenia <25,000/mm3 if associated with a bleeding event which does not result in hemodynamic instability but requires an elective platelet transfusion, or a life-threatening bleeding event which results in urgent intervention.
Time Frame: 3 weeks for Arm A; First cycle (Arm B - 3 weeks and Arm C- 4 weeks)
Population: 16/37 participants were not analyzed. 3 participants did not complete Cycle 1 and were replaced, and according to the protocol, DLTs were to be assessed in the first 6 participants. If 0 or 1 DLT occurred, treatment would continue at that dose for the remaining participants. Since only 1 DLT was observed in the first 6 participants, the dose was deemed acceptable, and the remaining 13 participants were treated at the same dose without further DLT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 10 | 5 | 6
Participants
  Grade 3 Rash maculopapular | 0 | 0 | 1
  Grade 4 Platelet count decreased | 0 | 1 | 0
  Grade 5 Death related to adverse event | 0 | 0 | 0

4. Secondary Outcome: Proportion of Grade 3 and/or Grade 4 Adverse Events
Description: Safety of the agent will be assessed by determining the grade of adverse events noted in each participant and reporting the fraction with grade 3 and/or grade 4 adverse events. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: Document adverse events from the first study intervention through 30 days after the participant received the last study treatment administration, approximately 30-353 days
Measure: Number; unit: Proportion of adverse events
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 13 | 5 | 19
Proportion of adverse events
  Grade 3 | 0.149 | 0.246 | 0.1191
  Grade 4 | 0.01 | 0.03 | 0.0255

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. PFS will begin at the on-study date and will consider progressions as well as death without progression as an event. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. PFS was measured using the Kaplan-Meier method and is reported along with a 95% confidence interval.
Time Frame: At 6 months
Population: 7/37 participants were not analyzed because 7 participants were not evaluable for response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 10 | 5 | 15
Months | 2.31 [1.38 to 6.5] | 1.44 [1.11 to 2.03] | 2.03 [1.84 to 5.79]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented using the Kaplan-Meier method and reported along with a 95% confidence interval. Response is measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response is disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: At 6 months
Population: 33/37 participants evaluable for CR/PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 1 | 0 | 3
Months | 3.71 [NA to NA] — A 95% confidence interval cannot be calculated from just one observation because there is no way to estimate variability or the spread of the data. |  | 16.67 [3.91 to 17.11]

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the date of on-study to the date of death from any cause or last follow up. OS was measured using the Kaplan-Meier method and is reported along with a 95% confidence interval.
Time Frame: maximum of 67.14 months
Population: 7/37 participants were not analyzed because 7 participants were not evaluable for response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 10 | 5 | 15
Months | 4.58 [2.13 to 12.78] | 2.89 [1.87 to 5.88] | 8.86 [2.95 to 17.31]

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events was monitored/assessed from the first study intervention through 30 days after the participant received last study treatment administration, 30 - 467 days or an average of 112.4 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
Number analyzed (Participants) | 13 | 5 | 19
Participants | 13 | 5 | 19

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed an average of 7.56 months. Adverse Events was monitored/assessed from the first study intervention through 30 days after the participant received last study treatment administration, 30 - 467 days or an average of 112.4 days.
Arm/Group | Arm A/M7824 (MSB0011359C) Monotherapy | Arm B/M7824 (MSB0011359C) Plus Topotecan | Arm C/M7824 (MSB0011359C) Plus Temozolomide
All-Cause Mortality (participants affected / at risk) | 13/13 | 5/5 | 18/19
Serious Adverse Events (participants affected / at risk) | 8/13 | 1/5 | 12/19
Other Adverse Events (participants affected / at risk) | 13/13 | 5/5 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A/M7824 (MSB0011359C) Monotherapy (N=13) | Arm B/M7824 (MSB0011359C) Plus Topotecan (N=5) | Arm C/M7824 (MSB0011359C) Plus Temozolomide (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 4 (4) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify: enteric neuropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify: Mucosal bleeding (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify: Altered mental status (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A/M7824 (MSB0011359C) Monotherapy (N=13) | Arm B/M7824 (MSB0011359C) Plus Topotecan (N=5) | Arm C/M7824 (MSB0011359C) Plus Temozolomide (N=19)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 0 (0) | 6 (6)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (6) | 1 (2) | 5 (12)
Alkaline phosphatase increased (Investigations) | 2 (6) | 1 (2) | 3 (6)
Anemia (Blood and lymphatic system disorders) | 7 (15) | 5 (7) | 10 (28)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 8 (12)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 1 (2) | 6 (14)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 4 (4)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1) | 3 (4)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
CPK increased (Investigations) | 0 (0) | 0 (0) | 2 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 2 (3) | 0 (0) | 3 (5)
Constipation (Gastrointestinal disorders) | 6 (6) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 2 (2)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 0 (0) | 8 (10)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 0 (0) | 5 (5)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1)
Eye disorders - Other, specify: Double vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify: Scotoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (7) | 1 (1) | 10 (14)
Fever (General disorders) | 1 (1) | 0 (0) | 4 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1) | 1 (15)
Gait disturbance (General disorders) | 2 (3) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Abdominal lump (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: Gum bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify: Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: abdominal pressure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify: broken tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify: Cervical lymph node (General disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify: poor quality of life (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 6 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 8 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (6)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (5) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Infections and infestations - Other, specify: Poison Ivy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify: c diff (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify: Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify: nasal contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (7) | 0 (0) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 1 (1) | 2 (3)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (12) | 1 (1) | 11 (27)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (12) | 2 (3) | 13 (19)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (3)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 4 (4)
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (5) | 4 (13) | 9 (28)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0) | 6 (12)
Psychiatric disorders - Other, specify: Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (9) | 0 (0) | 6 (14)
Renal and urinary disorders - Other, specify: Nocturia (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify: Hemoptysis - intermittent (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify: Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify: hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify: Keratoacanthomas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Keratocanthoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Scalp irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: actinic keratoses (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: actinic keratoses (Left thigh) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thyroid stimulating hormone increased (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Vascular disorders - Other, specify: Petechiae (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (9) | 1 (2) | 10 (17)
Weight loss (Investigations) | 3 (5) | 0 (0) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (3) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03554473/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03554473/ICF_001.pdf